CLINICAL TRIAL: NCT01868243
Title: Dabigatran Versus Warfarin After Mitral and Aortic Bioprosthesis Replacement for the Management of Atrial Fibrillation Postoperatively: Pilot Study
Brief Title: Dabigatran Versus Warfarin After Mitral and/or Aortic Bioprosthesis Replacement and Atrial Fibrillation Postoperatively
Acronym: DAWA
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: because a significant decrease of viable candidates for the study.
Sponsor: Hospital Ana Nery (Other)
Responsible Party: Principal Investigator, Andre Duraes, PhD, Andre Rodrigues Duraes, Hospital Ana Nery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAWA2013
Record Dates: First submitted 2013-05-28; First posted 2013-06-04 (Estimated); Results first posted 2015-10-09 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-09

CONDITIONS: Primary Disease
Keywords: Atrial Fibrillation; Bioprosthesis; Stroke; Dabigatran; Warfarin
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Dabigatran; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dabigatran (Experimental): Dabigatran 110 mg BID
  Interventions: Drug: Dabigatran
- Warfarin (Active Comparator): Warfarin adjusted-dose
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Dabigatran — Group 1 - Dabigatran 110 mg (50 patients)
  Other Names: Pradaxa® (dabigatran etexilate) 110mg twice daily
  Arms: Dabigatran
Drug: Warfarin — Warfarin adjusted-dose
  Other Names: Warfarin adjusted-dose
  Arms: Warfarin

SUMMARY:
DAWA is a phase 2, prospective, open-label, randomized, pilot study. The main variable to be observed in this study is intracardiac thrombus. There are no formal primary or secondary clinical efﬁcacy or safety outcomes because it is a pilot study.

DETAILED DESCRIPTION:
Mortality and morbidity events (reversible ischemic neurological deficit, ischemic and hemorrhagic stroke, systemic embolism, any bleeding, prosthesis valve thrombosis and death) were evaluated in an exploratory manner. The details of the trial design have been previously described.8 The trial protocol was approved by the local ethics and research committee in the city of Salvador-Brazil, and written informed consent was obtained from all patients. An independent data and safety monitoring board closely monitored the trial. All the members contributed to the interpretation of the results, wrote the first version of the manuscript and approved all versions, made the decision to submit the manuscript for publication, and vouch for the accuracy and completeness of the data reported and the fidelity of this article to the study protocol.

Patients eligible for inclusion in the study were 18 to 64 years old, underwent mitral and/or aortic bioprosthesis valve replacement at least 3 months prior to entering the study and had documented AF postoperatively in addition to exclusion of atrial thrombus or valve prosthesis thrombosis by transesophageal echocardiography (TEE). Non-contrast brain computed tomography (CT) without hemorrhage or findings of acute cerebral infarction on the last 2 days of screening was also necessary.

Patients were randomly assigned to receive dabigatran or warfarin by a computer generated list of random numbers performed to 1:1 ratio between the groups. Following that, the allocation sequence was concealed from the researcher enrolling participants in sequentially numbered, opaque, black, sealed envelopes. After randomization, patients had study visits scheduled at 7 days (via telephone) and at 30 days (personally) with a monthly follow-up for 90 days. After this, non-contrast brain CT and TEE were repeated. The former was executed to document possible cerebral events with no clinical expression and the latter to analyze the incidence of intracardiac thrombi, new dense spontaneous echo contrast (SEC) or its resolution, in addition to thrombosis or dysfunction of valvular prosthesis.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 64 years at entry
2. Patients with mitral and/or aorthic valve bioprosthesis for at least 3 months postoperatively
3. There is 12-lead electrocardiogram documented AF on the day of screening or randomization; or a 24-hour Holter electrocardiogram recording showing AF episodes postoperatively
4. Brain computed tomography scan without hemorrhage or findings of acute cerebral infarction on the last 2 days of screening
5. Exclusion of atrial thrombus or valve prosthesis thrombosis by transesophageal echocardiograph on the last 2 days of screening
6. Written, informed consent

Exclusion Criteria:

1. Previous hemorrhagic stroke
2. Ischemic stroke in the last 6 months
3. Severe renal impairment (creatinine clearance rates < 30 ml/min)
4. Active liver disease (any etiology)
5. Concomitant use of any antiplatelet (aspirin, clopidogrel, prasugrel, ticagrelor, ticlopidine, etc)
6. Increased risk of bleeding (congenital or acquired)
7. Uncontrolled hypertension
8. Gastrointestinal hemorrhage within the past year
9. Anemia (hemoglobin level <10 g/dL) or thrombocytopenia (platelet count < 100 × 109/L)
10. Active infective endocarditis
11. Pregnant or lactating women

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2013-08; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andre R Duraes, Professor, Principal Investigator — Hospital Ana Nery
Locations (1):
- Hospital Ana Nery, Salvador, Estado de Bahia, Brazil

REFERENCES:
- [Background] Nkomo VT, Gardin JM, Skelton TN, Gottdiener JS, Scott CG, Enriquez-Sarano M. Burden of valvular heart diseases: a population-based study. Lancet. 2006 Sep 16;368(9540):1005-11. doi: 10.1016/S0140-6736(06)69208-8. PMID 16980116
- [Background] Carapetis JR, Steer AC, Mulholland EK, Weber M. The global burden of group A streptococcal diseases. Lancet Infect Dis. 2005 Nov;5(11):685-94. doi: 10.1016/S1473-3099(05)70267-X. PMID 16253886
- [Background] Sun JC, Davidson MJ, Lamy A, Eikelboom JW. Antithrombotic management of patients with prosthetic heart valves: current evidence and future trends. Lancet. 2009 Aug 15;374(9689):565-76. doi: 10.1016/S0140-6736(09)60780-7. PMID 19683642
- [Background] Heras M, Chesebro JH, Fuster V, Penny WJ, Grill DE, Bailey KR, Danielson GK, Orszulak TA, Pluth JR, Puga FJ, et al. High risk of thromboemboli early after bioprosthetic cardiac valve replacement. J Am Coll Cardiol. 1995 Apr;25(5):1111-9. doi: 10.1016/0735-1097(94)00563-6. PMID 7897124
- [Background] Connolly SJ, Ezekowitz MD, Yusuf S, Eikelboom J, Oldgren J, Parekh A, Pogue J, Reilly PA, Themeles E, Varrone J, Wang S, Alings M, Xavier D, Zhu J, Diaz R, Lewis BS, Darius H, Diener HC, Joyner CD, Wallentin L; RE-LY Steering Committee and Investigators. Dabigatran versus warfarin in patients with atrial fibrillation. N Engl J Med. 2009 Sep 17;361(12):1139-51. doi: 10.1056/NEJMoa0905561. Epub 2009 Aug 30. PMID 19717844
- [Derived] Duraes AR, de Souza Roriz P, de Almeida Nunes B, Albuquerque FP, de Bulhoes FV, de Souza Fernandes AM, Aras R. Dabigatran Versus Warfarin After Bioprosthesis Valve Replacement for the Management of Atrial Fibrillation Postoperatively: DAWA Pilot Study. Drugs R D. 2016 Jun;16(2):149-54. doi: 10.1007/s40268-016-0124-1. PMID 26892845
- [Derived] Duraes AR, Roriz PD, Bulhoes FV, Nunes BD, Muniz JQ, Neto IN, Fernandes AM, Reis FJ, Camara EJ, Junior ED, Segundo DTs, Silva FP, Aras R. Dabigatran versus warfarin after bioprosthesis valve replacement for the management of atrial fibrillation postoperatively: protocol. JMIR Res Protoc. 2014 Apr 1;3(2):e21. doi: 10.2196/resprot.3014. PMID 24691436

RESULTS

PARTICIPANT FLOW:
Groups:
- Dabigatran: Dabigatran 110 mg BID
  Dabigatran: Group 1 - Dabigatran 110 mg
- Warfarin: Warfarin adjusted-dose
  Warfarin: Warfarin adjusted-dose (INR 2.0-3.0)
Period: Overall Study
Arm/Group | Dabigatran | Warfarin
Started | 15 | 12
Completed | 15 | 11
Not Completed | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dabigatran | Warfarin | Total
Number analyzed (Participants) | 15 | 12 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (10) | 46 (6) | 47 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  Brazil | 15 | 12 | 27

OUTCOME MEASURES:

1. Primary Outcome: Intracardiac Thrombus
Description: The primary endpoint was the detection of intracardiac thrombus in TEE at the end of follow-up (90 days).
Time Frame: 90 days
Population: A total of 34 patients were selected between August 2013 and November 2014 (6 were excluded for previous intracardiac thrombus; 1 for unstable INR control). Of the 27 randomized, 15 were assigned to receive dabigatran and 12 to receive warfarin.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 15 | 12
participants | 0 [0 to 0] | 1 [0.9 to 1.3]

2. Secondary Outcome: Spontaneous Echo Contrast
Description: Spontaneous Echo Contrast showed in Transesophageal echocardiography
Time Frame: 90 days
Measure: Number; unit: participants
Arm/Group | Dabigatran | Warfarin
Number analyzed (Participants) | 15 | 12
participants | 2 | 1

ADVERSE EVENTS:
Arm/Group | Dabigatran | Warfarin
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/12
Other Adverse Events (participants affected / at risk) | 1/15 | 1/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dabigatran (N=15) | Warfarin (N=12)
Stroke (Nervous system disorders) | 1 (1) | 0 (0) — Ischemic Stroke
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dabigatran (N=15) | Warfarin (N=12)
Bleeding (Gastrointestinal disorders) | 1 (1) | 1 (1) — Gastrointestinal bleeding

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No